CLINICAL TRIAL: NCT01914874
Title: Efficacy of an Enhanced Mindfulness-based Intervention for Social Anxiety Disorder: A Pilot Feasibility Randomized Controlled Trial
Brief Title: Efficacy of a Mindfulness Meditation Program for Social Anxiety Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Montfort (Other)
Responsible Party: Principal Investigator, Diana Koszycki, Research Chair In Mental Health/Senior Scientist, Hopital Montfort
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DK-05-02-13
Record Dates: First submitted 2013-07-30; First posted 2013-08-02 (Estimated); Last update posted 2015-07-01 (Estimated); Status verified 2015-06

CONDITIONS: Social Anxiety Disorder
Keywords: Community Sample
MeSH Terms: conditions — Phobia, Social | interventions — Mindfulness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mindfulness Meditation (Experimental): 12 weekly sessions in group format
  Interventions: Behavioral: Mindfulness Meditation
- Wait-list (No Intervention): Patients will receive the mindfulness intervention after a 12-week wait period

INTERVENTIONS:
Behavioral: Mindfulness Meditation
  Arms: Mindfulness Meditation

SUMMARY:
The aim of this study is to evaluate the feasibility and initial efficacy of an enhanced mindfulness-based program that includes "mindful exposure" to reduce anxiety and avoidance of social situations, and the Buddhist practice of self-compassion aimed at reducing harsh judgment and self-criticism that is characteristic of people with social anxiety disorder.

DETAILED DESCRIPTION:
The purpose of this pilot study is to evaluate the feasibility and initial efficacy of an enhanced mindfulness-based intervention for SAD (MIND-SAD) that incorporates the following components: training in classical mindfulness, including concentration and insight (vipassana) meditation; training in self-compassion; and mindful exposure. An exploratory aim of the study is to evaluate the effects of the mindfulness intervention on biological markers of stress reactivity, including salivary cortisoland salivary alpha-amylase. The study is a two-arm, parallel design, prospective study comparing 12 weekly sessions of MIND-SAD delivered in a group format versus a wait-list control (WLC).

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of Social Anxiety Disorder; Baseline score of 30 or higher on the Liebowitz Social Anxiety Scale; Baseline score of 4 or higher on the Clinical Global Impression of Severity

Exclusion Criteria:

* Lifetime history of psychosis or bipolar disorder; substance abuse in the past 12 months; diagnosis of borderline or antisocial personality disorder; serious suicide risk; currently in psychotherapy; regular meditation or yoga practice in the past 12 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2013-07; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Clinician-rated Liebowitz Social Phobia Scale | change from baseline at weeks 6, 12 and 3 months follow-up
Social Phobia Inventory | change from baseline at weeks 6, 12 and 3 months follow-up

SECONDARY OUTCOMES:
Beck Depression Inventory | change from baseline at weeks 6, 12 and 3 months follow-up
Social Adjustment Scale-Self-Report | change from baseline at weeks 6 and 12 and 3 months follow-up
CGI-Severity of Illness | change from baseline at weeks 6, 12 and 3 months follow-up
Self-Compassion Scale | change from baseline at weeks 6, 12 and 3-months follow-up
Five Facet Mindfulness Questionnaire | change from baseline at weeks 6, 12 and 3 months follow-up

OTHER OUTCOMES:
Study compliance: attendance and homework | compliance will be assessed at each week during the 12-week mndfulness meditation program
Salivary cortisol | change from baseline at week 12
Salivary alpha-amylase | change from baseline at week 12

CONTACTS AND LOCATIONS:
Overall Officials: Diana Koszycki, PhD, Principal Investigator — Montfort Hospital and University of Ottawa
Locations (1):
- Montfort Hospital, Ottawa, Ontario, Canada